CLINICAL TRIAL: NCT04980547
Title: Evaluation of the Surgical Proficiency and Effectiveness of the Acumed(R) Scapholunate Repair System in Primary Scapholunate Instability Among Canadians
Brief Title: Evaluation of the Surgical Proficiency and Effectiveness of the Acumed Scapholunate Repair System in Primary Scapholunate Instability Among Canadians
Acronym: CanRASL
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Collaborators: Acumed, LLC (Industry)
Responsible Party: Principal Investigator, Neil White, Clinical Assistant Professor, Section of Orthopaedics, Hand & Wrist Surgeon, University of Calgary, University of Calgary
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB20-2245
Record Dates: First submitted 2021-07-15; First posted 2021-07-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Complete Tear of Scapholunate Ligament; Scapholunate Dissociation
Keywords: Scapholunate interosseous ligament; Reduction and association of the scaphoid and lunate; RASL; Acumed Scapholunate Repair System

STUDY DESIGN:
Intervention Model Description: This is a prospective, multi-centre, non-randomized, and non-blinded follow-up study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- ACUMED® Scapholunate Repair System (Experimental): All participants in this trial will undergo the surgical RASL procedure using the ACUMED® Scapholunate Repair System.
  Interventions: Device: ACUMED® Scapholunate Repair System Group

INTERVENTIONS:
Device: ACUMED® Scapholunate Repair System Group — To address the technical difficulties associated with the RASL procedure, Dr. Mel Rosenwasser developed an external over-the-top jig that in theory enables accurate and easy scapholunate-axis screw placement. The Acumed Scapholunate Repair System was designed treat patients with acute or chronic, static or dynamic scapholunate instability in the absence of significant capitolunate osteoarthritis, scapholunate ligament repair, scapholunate reduction, lunotriquetral ligament repair, lunotriquetral reduction, and carpal instability. This new Scapholunate Repair System features a targeting guide designed to enable the surgeon to reproducibly place the implant in optimal position. The implant allows physiologic intercarpal scapholunate rotation by means of a free rotation design. The procedure can forestall progressive osteoarthritis and the need for secondary salvage procedures.

SUMMARY:
This study is a prospective, multi-centre, non-randomized, and non-blinded follow-up study to assess the efficacy and effectiveness of the ACUMED® Scapholunate Repair System in primary scapholunate interosseous ligament (SLIL) reconstruction.

DETAILED DESCRIPTION:
The scapholunate interosseous ligament (SLIL) of the wrist can be likened to the ACL of the knee as an often-injured ligament causing joint instability that frequently impairs function and requires surgical reconstruction. Yet wrist surgeons are significantly behind knee surgeons in their ability to achieve consistent and reliable outcomes with surgical reconstruction of this ligament. This ligament is often treated using a surgical procedure of reduction and association of scaphoid and lunate (RASL). However, this procedure is accompanied with technical challenges regarding proper screw placement and trajectory.

The ACUMED® Scapholunate Repair System presents as a novel and innovated device that has the potential to improve surgeon proficiency with the RASL procedure. The purpose of this trial is to assess the efficacy and effectiveness of the ACUMED® Scapholunate Repair System in primary scapholunate interosseous ligament (SLIL) reconstruction. The study will assess the surgeon learning curve with the ACUMED® Scapholunate Repair System, record safety, complications, outcomes and adverse events for 2 years after surgery. This study will generate clinical evidence to support and maintain product registration in global markets.

Patients presenting with sub-acute or chronic (>8 weeks) primary SLIL instability that will be treated surgically at up to 20 study sites across Canada. A total of 50 wrists will be enrolled into the study and surgeons will utilize the ACUMED® Scapholunate Repair System during the surgical procedure. The study is expected to enroll all subjects within a 2-year time frame, and patients will be followed for 2 years after surgery. Subjects for whom the informed consent process has been completed and have been implanted with the study product will be considered enrolled.

At baseline, research staff will obtain data regarding participant demographics, injury characteristics, and medical history. Pre-operatively, participants will also be assessed for range of motion and grip strength and will have completed radiographs and three wrist function questionnaires, the DASH, the PRWE, and the PROMIS. Surgeons will answer questionnaires at the start of the study, after each surgical case, and at the end of the study to provide an assessment of the repair system's utility. The quality of screw placement will be graded on a newly created scale (from retrospective chart review of prior RASL procedures) to measure screw trajectory and final placement. Participants will have follow standard of care follow up timeline with preoperative visits at 2-, 8-, 12, 24- weeks, 1 year, 18 months, and 2 years. At each follow up visit, range of motion data, grip strength (after 24 weeks), and questionnaires will be completed.

Data will be reported as numbers and percentages of total for categorical data, and as mean and standard deviation of the mean with 95% confidence intervals for continuous variables. Ordinal data from the Likert scale surgeon questionnaire and screw placement grading scales will also be analyzed using parametric statistics (1, 2). Total scores from the scale items will be analyzed using the Kappa statistics. Independent sample t-tests will be used to compare the mean DASH, PRWE and PROMIS scores and for time to return to work, school, and sports. For secondary analysis, an analysis of variance will be completed for the DASH, PRWE and PROMIS scores, range of motion data and grip strength at each follow-up time interval.

ELIGIBILITY:
Inclusion Criteria:

* Subject has primary, chronic (> 6 weeks) scapholunate instability diagnosed by X-ray, dynamic X-ray, MRI/MRI arthrogram and/or arthroscopy
* Subject is a suitable candidate for RASL repair with the ACUMED® Scapholunate Repair System
* Subject is willing and able to participate in required follow-up visits and can complete study activities.
* Subject provides informed consent

Exclusion Criteria:

* Subject has scapholunate advanced collapse wrist arthritis above grade I (styloid only)
* Subject has conditions that would eliminate or tend to eliminate adequate implant support:

  1. Blood supply limitations;
  2. Insufficient quantity or quality of bone support (osteoporosis, metabolic disorders which may impair bone formation, tumor, osteomalacia, etc.).
* Subject has mental or neurological conditions which impair their ability or willingness to restrict activities that may put the affected limb at risk.
* Subject has physical conditions that tend to place extreme loads on the implants (Charcot joints, muscle deficiencies etc.).
* Subject has neuromuscular dysfunctions (paralysis, myolysis, etc.) which could cause instability of the wrist after surgery
* Subject has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the study
* Subject has an active infection - systemic or at the site of intended surgery
* Subject has a known allergy to any component of the devices used in the study
* Subject is pregnant or breast feeding
* Subject is entered in another investigational drug, biologic, or device study within 30 days of active study participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Assess surgical proficiencies and effectiveness with the ACUMED® Scapholunate Repair System | Immediately after surgery
  Surgeons will complete a standardized proprietary questionnaire at the start of the study and on a case by case basis following each surgical procedure (Post-operatively). The goal is to measure and track the level of surgeon comfort and proficiency with the ACUMED® Scapholunate Repair System. Surgical time, tourniquet time and fluoroscopy time will be used a surrogate measures of surgical proficiency.
Quality of Screw Placement | Immediately after surgery
  Scapholunate screw trajectory will be validated and graded based on screw angle (ideally 23 degrees), position in the ulnar vertex (proximal ulnar corner), and sagittal alignment (middle third of scaphoid) based on intra-operative or immediate post-operative AP and lateral X-rays.

SECONDARY OUTCOMES:
Correlate Clinical Outcomes to Reduction and Screw Trajectory | 2 years
  Functional outcomes will be assessed using the Patient-Rated Wrist Evaluation (PRWE), Disabilities of the Arm, Shoulder and Hand (DASH), PROMIS Upper Extremity, and Visual Analogue Pain Scale (VAS).
Report Safety Complications and Adverse Events | 2 years
  Complications, adverse events and serious adverse events possibly related, probably related, or related to the device and/or the surgical procedure that may adversely affect study functional outcome scores will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Neil J White, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geissler WB. Arthroscopically assisted reduction of intra-articular fractures of the distal radius. Hand Clin. 1995 Feb;11(1):19-29. PMID 7751327
- [Background] Messina JC, Van Overstraeten L, Luchetti R, Fairplay T, Mathoulin CL. The EWAS Classification of Scapholunate Tears: An Anatomical Arthroscopic Study. J Wrist Surg. 2013 May;2(2):105-9. doi: 10.1055/s-0033-1345265. PMID 24436801
- [Background] Montgomery SJ, Rollick NJ, Kubik JF, Meldrum AR, White NJ. Surgical outcomes of chronic isolated scapholunate interosseous ligament injuries: a systematic review of 805 wrists. Can J Surg. 2019 Mar 22;62(3):1-12. doi: 10.1503/cjs.006918. Online ahead of print. PMID 30900438
- See also: SCRUBS Research Group — http://www.scrubsresearch.com/